CLINICAL TRIAL: NCT00025688
Title: A Randomized, Phase II Trial of Weekly Taxol (Paclitaxel) Versus Weekly Taxol Plus Paraplatin (Carboplatin) as First-Line Chemotherapy in Patients Age 65 Years or Older With Metastatic Breast Cancer
Brief Title: Paclitaxel With or Without Carboplatin in Treating Women With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068992; THERADEX-B00-1370; BMS-TAX/MEN.13
Record Dates: First submitted 2001-10-11; First posted 2003-08-05 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2006-09

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if paclitaxel is more effective with or without carboplatin in treating stage IV breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of paclitaxel with or without carboplatin in treating women who have stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the objective response rate in women treated with paclitaxel with or without carboplatin as first-line chemotherapy for metastatic breast cancer.
* Compare the overall survival, time to disease progression, and duration of response in these patients treated with these regimens.
* Compare the safety of these regimens in this patient population.
* Compare the quality of life of these patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior adjuvant chemotherapy (yes vs no) and ECOG performance status (0-1 vs 2). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive paclitaxel IV over 1 hour weekly for 3 weeks.
* Arm II:Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes weekly for 3 weeks.

Treatment in both arms continues every 4 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, before each course during study, and then after completion of study.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 220 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Must have clinical evidence of stage IV (M1) disease
* HER-2/neu negative (0, 1+, or 2+ by immunohistochemistry or fluorescent in situ hybridization) OR status unknown
* At least 1 measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Patients with bone-only disease are not eligible
* Ineligible if currently experiencing a complete or partial response to prior hormonal therapy
* Patients with disease progression after prior response to hormonal therapy are eligible
* Disease progression without prior hormonal therapy is allowed
* Stable or asymptomatic brain metastasis allowed if:

  * Other measurable disease exists
  * Cranial irradiation completed and brain metastasis stable for at least 4 weeks before study
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Pre- or post-menopausal

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2 times ULN

Renal:

* Creatinine no greater than 2 times ULN
* Corrected calcium less than 12 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No documented myocardial infarction within the past 6 months
* No congestive heart failure
* No unstable angina
* No clinically significant pericardial effusion or arrhythmia

Other:

* No active serious infection
* No prior significant allergic reactions to drugs containing Cremophor, such as teniposide, cyclosporine, or vitamin K
* No clinically significant (greater than grade 1) peripheral neuropathy
* No other serious underlying medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 6 months since prior adjuvant bone marrow or peripheral blood stem cell transplantation
* More than 6 months since prior adjuvant monoclonal antibody therapy
* More than 6 months since prior adjuvant vaccine therapy
* No prior trastuzumab (Herceptin)
* No concurrent anticancer immunotherapy

Chemotherapy:

* No prior chemotherapy for metastatic breast cancer
* More than 6 months since prior adjuvant high-dose chemotherapy
* More than 6 months since prior adjuvant taxanes or any other adjuvant chemotherapy
* Prior adjuvant taxanes allowed only if administered every 3 weeks

Endocrine therapy:

* See Disease Characteristics
* Any number of prior hormonal therapies for metastatic breast cancer allowed

  * Patients with definite signs of progression may begin study therapy immediately after stopping hormonal therapy
* No concurrent anticancer hormonal agents (including megestrol)

Radiotherapy:

* At least 3 weeks since prior radiotherapy (4 weeks for cranial irradiation)
* No prior radiotherapy to 30% or more of bone marrow
* No concurrent radiotherapy except for palliation of painful bone metastasis or pathologic fractures to the area of known lytic disease

Surgery:

* At least 3 weeks since prior major surgery

Other:

* More than 6 months since prior neoadjuvant therapy
* No other concurrent anticancer drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic
Locations (25):
- United States (25):
  - Highlands Oncology Group, Springdale, Arkansas
  - Monterey Bay Oncology, Monterey, California
  - Wilshire Oncology Medical Group, Inc., Pomona, California
  - University of California Davis Cancer Center, Sacramento, California
  - New Britain General Hospital, New Britain, Connecticut
  - Center for Hematology and Oncology, Boca Raton, Florida
  - Cancer Research Network, Inc., Hollywood, Florida
  - Mayo Clinic, Jacksonville, Florida
  - MacNeal Cancer Center, Berwyn, Illinois
  - Oncology Specialists, SC, Park Ridge, Illinois
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Maryland Hematology/Oncology Associates, Baltimore, Maryland
  - St. John's Mercy Medical Center, St Louis, Missouri
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Finger Lakes Community Cancer Center, Clifton Springs, New York
  - Clinical Hematology & Oncology Service, Inc., Akron, Ohio
  - Scranton Hematology-Oncology, Scranton, Pennsylvania
  - East Tennessee Oncology/Hematology, P.C., Knoxville, Tennessee
  - West Clinic, Memphis, Tennessee
  - Texas Cancer Care, Fort Worth, Texas
  - Oncology Consultants, Houston, Texas
  - Scott and White Clinic, Temple, Texas
  - Northern Virginia Oncology Group, P.C., Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Dean Medical Center, Madison, Wisconsin